CLINICAL TRIAL: NCT05301205
Title: Perioperative Administration of Gabapentin for Reducing Inhalational Anesthetic Consumption
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Samir Wahdan, Lecturer of Anesthesia, Pain management and Surgical ICU, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N-48-2021
Record Dates: First submitted 2022-03-19; First posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Gabapentin
MeSH Terms: interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group I (Active Comparator): will be received oral gabapentin capsule 1200 mg 2h pre-operatively.
  Interventions: Drug: oral gabapentin
- group II (Active Comparator): will be received oral gabapentin capsule 600 mg 2h pre-operatively.
  Interventions: Drug: oral gabapentin
- Group III (No Intervention): will be received placebo capsules at 2 hours preoperatively.

INTERVENTIONS:
Drug: oral gabapentin — will be received oral gabapentin capsule 2 HOURS pre-operatively.
  Arms: group I; group II

SUMMARY:
Gabapentin, a structural analog of gamma aminobutyric acid (GABA), was introduced within the us as an anticonvulsant, used clinically to treat epilepsy. The drug causes amino acids release within the medulla spinalis dorsal horn and thus decreasing response to neural inputs and stabilizing the nervous activity. The mechanism of action of gabapentin on neuropathic pain is assumed to bind to the alpha 2 delta subunit of the voltage-dependent calcium channel within the central systema nervosum , reducing calcium influx into the nerve terminals and decreases the release of neurotransmitters like glutamate . Gabapentin, therefore, can be used for controlling chronic pain, as in diabetic neuropathy and other neuropathic disorders . Some studies examined the effectiveness of gabapentin for acute postoperative pain management for gynecological surgery, lumbar spinal surgery, arthroplasty, and thoracic surgery . A recent study concluded that gabapentin has a role in preoperative anxiolysis, attenuation of hemodynamic response to intubation, prevention of postoperative nausea and vomiting (PONV) and finally postoperative delirium . Up to date, the effect of preoperative gabapentin on inhaled anesthetic depth is unknown

ELIGIBILITY:
1. Inclusion criteria:

   * Patients aged from 18 to 60 years.
   * ASA I-II.
   * Undergoing craniotomy for intracranial tumors.
2. Exclusion criteria:

   * Patient refusal
   * Patients younger than 18 or above 60 years old
   * patients with (ASA) physical status ≥ III
   * patients with compromised cardiovascular, renal, hepatic or neurological function
   * Known allergy to study drug.
   * Contraindication or chronic use (consistent use for longer than 3 months) to any of the study drugs
   * Suffered from severe psychiatric disease or drug addiction;
   * History of parenteral or oral analgesic intake within the last 48hours

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 96 (Estimated)
Dates: Start 2021-06-25 (Actual); Primary Completion 2023-06-13 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
sevoflurane consumption | 4 hours
  Intra-operative consumption of sevoflurane will be measured and recorded (ml/hr).

SECONDARY OUTCOMES:
nalbuphine consumption | 24 hours
  postoperative nalbuphine consumption by mg
Intraoperative fentanyl consumption. | 6 hours
  Intraoperative fentanyl consumption by mic

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
still working